CLINICAL TRIAL: NCT01997801
Title: The Efficacy of Intraoperative Ketamine in Patients Undergoing Robot-assisted Thyroidectomy
Brief Title: Ketamine in Robot-assisted Thyroidectomy
Acronym: KEThyRobot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Pyoung Park, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SNUH_KEThyRobot
Record Dates: First submitted 2013-11-18; First posted 2013-11-28 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Thyroid; Acute Pain; Chronic Pain
Keywords: Thyroidectomy; Endoscopy; Ketamine; Acute Pain; Chronic Pain; Postoperative period
MeSH Terms: conditions — Thyroid Diseases; Acute Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- C group (Placebo Comparator): In C group, NS infusion will be done intraoperatively.
  Interventions: Drug: NS infusion
- KET group (Experimental): In KET group, ketamine infusion will be done intraoperatively(0.25 mg/kg bolus injection following 100 mcg/kg/hr till the end of surgery).
  Interventions: Drug: Ketamine infusion

INTERVENTIONS:
Drug: Ketamine infusion — Ketamine will be infused intraoperatively (0.25 mg/kg intravenous bolus following continuous infusion of 100 mcg/kg/hr).
  Arms: KET group
Drug: NS infusion — Normal saline will be infused intraoperatively.
  Arms: C group

SUMMARY:
In this prospective double-blinded study, The investigators compared acute postoperative pain and rescue analgesic demand during postoperative period after robot thyroidectomy between ketamine and placebo groups.

DETAILED DESCRIPTION:
Robot-assisted endoscopic thyroidectomy has been popularized due to cosmetic advantages. Despite small incisions, robot thyroidectomy did not offer satisfactory reduction in postoperative pain compared to open thyroidectomy. Ketamine is a non-competitive N-methyl-D-aspartate (NMDA) receptor blocker and takes some attractive advantages in terms of pain control. When low dose ketamine is perioperatively administrated, opioid sparing effect during postoperative period is reported in various surgical procedures such as spine, thoracic, and gynecologic surgery. Ketamine's beneficial effect on postoperative pain has not been investigated in patients undergoing robot thyroidectomy. The investigators hypothesized that perioperative ketamine administration can reduce acute postoperative pain after robot thyroidectomy and the incidence of chronic pain hypoesthesia on anterior chest at 3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for robot-assisted thyroidectomy
* ASA I-III

Exclusion Criteria:

* Patients with renal dysfunction
* Patients with hepatic dysfunction
* Patients with neurologic dysfunction
* Patients with the history of drug addiction
* Patients with chronic pain
* Patients who are allergic to ketamine
* Patients with increased ocular or intracranial pressure
* Patients with the risk of aspiration

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Pain at 24 hour postoperatively | at 24 hour postoperatively
  Pain at 24 hour postoperatively will be evaluates using 11 point scale (0:no pain, 10:worst imaginable)

SECONDARY OUTCOMES:
Pain at 3, 6, 12, 48 and 72 hour postoperatively | at 3, 6, 12, 48 and 72 hour postoperatively
  Pain at 3, 6, 12, 48 and 72 hour postoperatively will be evaluated using 11-point scale 0:no pain, 10:worst imaginable)
Time to the first analgesics postoperatively | At 24 hours postoperatively
  Time from the end of anesthesia till the first analgesic agent will be recorded at 24 hours postoperatively.
Analgesic requirements for 24 hours after surgery | at 24 hours postoperatively
  Analgesic requirements for 24 hours after surgery will be evaluated.
Chronic pain at 3 month after surgery | At 3 month after surgery
  Chronic pain at 3 month after surgery will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Pyoung Park, PhD, Study Director — Seoul National University of Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee J, Park HP, Jeong MH, Son JD, Kim HC. Efficacy of ketamine for postoperative pain following robotic thyroidectomy: A prospective randomised study. J Int Med Res. 2018 Mar;46(3):1109-1120. doi: 10.1177/0300060517734679. Epub 2017 Nov 10. PMID 29124992